CLINICAL TRIAL: NCT04544163
Title: Magnesium Versus High Dose Fentanyl in Attenuating Stress Response to Endotracheal Intubation
Brief Title: Magnesium Versus High Dose Fentanyl in Endotracheal Intubation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Cancer Institute, Egypt (Other)
Responsible Party: Principal Investigator, Walaa Youssef Elsabeeny, Lecturer of anesthesia and pain management, National Cancer Institute, Egypt
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AP2007-50108
Record Dates: First submitted 2020-09-03; First posted 2020-09-10 (Actual); Last update posted 2021-05-11 (Actual); Status verified 2021-05

CONDITIONS: Stress Response
MeSH Terms: conditions — Fractures, Stress | interventions — Fentanyl; Lidocaine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Magnesium sulphate- Fentanyl (Experimental): 30 mg per kg MgSo4 infusion in 100 ml saline over 10 minutes
  Interventions: Drug: Magnesium sulfate- Fentanyl; Drug: Fentanyl 2Mcg/kg
- Fentanyl 4 mic (Experimental): 4 mic per kg fentanyl i.v
  Interventions: Drug: Fentanyl 4Mcg/kg
- Fentanyl (Active Comparator): 2 mic per kg fentanyl i.v
  Interventions: Drug: Fentanyl 2Mcg/kg
- Lidocaine- Fentanyl (Experimental): Lidocaine 1.5 mg/kg
  Interventions: Drug: Fentanyl 2Mcg/kg; Drug: Lidocaine 1.5 mg/kg

INTERVENTIONS:
Drug: Magnesium sulfate- Fentanyl — drug administration before intubation
  Other Names: MgSo4
  Arms: Magnesium sulphate- Fentanyl
Drug: Fentanyl 4Mcg/kg — drug administration with induction of anesthesia
  Other Names: high dose fentanyl
  Arms: Fentanyl 4 mic
Drug: Fentanyl 2Mcg/kg — drug administration with induction of anesthesia
  Other Names: Conventional anesthesia
  Arms: Fentanyl; Lidocaine- Fentanyl; Magnesium sulphate- Fentanyl
Drug: Lidocaine 1.5 mg/kg — drug administaration 90 sec before intubation
  Other Names: Lidocaine
  Arms: Lidocaine- Fentanyl

SUMMARY:
this study is designed to assess the efficacy of MgSO4 versus high dose fentanyl compared to conventional anesthesia in attenuating stress response to intubation

DETAILED DESCRIPTION:
to assess the effect of MgSO4 combined with fentanyl compared to high dose fentanyl in attenuating stress response in cancer patients undergoing surgeries under general anesthesia requiring endotracheal intubation

ELIGIBILITY:
Inclusion Criteria:

* Cancer patients undergoing surgery under general anesthesia requiring endotracheal intubation
* ASA I II
* 18 to 60

Exclusion Criteria:

* allergy to any of the used drugs
* renal or hepatic impairment
* hypertensive patients, patients with cardiovascular or cerebrovascular diseases

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 160 (Actual)
Dates: Start 2020-09-05 (Actual); Primary Completion 2021-05-02 (Actual); Study Completion 2021-05-05 (Actual)

PRIMARY OUTCOMES:
heart rate values | 5 minutes
  changes in heart rate values after intubation

SECONDARY OUTCOMES:
blood pressure | 5 minutes
  mean arterial blood pressure values
coughing during intubation | lntubation time
  coughing during intubation

CONTACTS AND LOCATIONS:
Overall Officials: Walaa Y Elsabeeny, MD, Principal Investigator — Lecturer; Nahla N Shehab, MD, Principal Investigator — Lecturer
Locations (1):
- Walaa Y Elsabeeny, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Yes
data will be available upon reasonable request through contacting the corresponding author